CLINICAL TRIAL: NCT02207218
Title: A Multicentre, Non-interventional Post Marketing Study of Safety and Efficacy of NovoEight® (rFVIII) During Long-Term Treatment of Haemophilia A in Japan
Brief Title: To Investigate Safety and Efficacy of NovoEight® (rFVIII) During Long-term Treatment of Haemophilia A in Japan
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN7008-4105; U1111-1144-8212 (Other: WHO)
Record Dates: First submitted 2014-08-01; First posted 2014-08-04 (Estimated); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII N8

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NovoEight®
  Interventions: Drug: turoctocog alfa

INTERVENTIONS:
Drug: turoctocog alfa — No treatment given. Patients will be treated with commercially available NovoEight®. Patients will be treated according to local clinical practice at the direction of the physician.

SUMMARY:
This study is conducted in Asia. The aim of this study is to evaluate the safety and efficacy of NovoEight® (recombinant factor VIII) in patients with haemophilia A in Japan in the setting of routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedure related to recording of data according to the protocol
* Male and female patients with the diagnosis of haemophilia A
* Age range is 0 year and above
* A decision to initiate treatment with commercially available NovoEight® has been made by the patient/parent and the physician

Exclusion Criteria:

* Known or suspected allergy to study product(s) or related products
* Previous participation in this study. Participation is defined as informed consent obtained
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: NovoEight® in prevention, treatment of bleeds and prevention of bleeds during and after surgery in previously treated patients (PTPs) and previously untreated patients (PUPs) with haemophilia A in routine clinical setting in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-08-04 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AEs) | Week 0- 104

SECONDARY OUTCOMES:
Frequency of Adverse Reactions (ARs) | Week 0- 104
Frequency of Serious Adverse Events (SAEs) | Week 0- 104
Frequency of Serious Adverse Reactions (SARs) | Week 0- 104
Haemostatic effect of NovoEight® in the treatment of bleeds according to a predefined four point scale: Excellent, Good, Moderate, or None for patients with preventive regimen and on-demand treatment regimen, respectively | Week 0- 104
Haemostatic effect of NovoEight® during surgical procedures assessed by evaluation according to a predefined four point scale: Excellent, Good, Moderate, or None | Week 0- 104
Annualised bleeding rate for patients using NovoEight® for preventive regimen | Week 0- 104
Total consumption of NovoEight® per patient (prevention, treatment of bleeds and surgery) per year (IU/kg BW/year/patient) | Week 0- 104
Consumption of NovoEight® per bleed (IU/kg BW/bleeding episode) | Week 0- 104
Consumption of NovoEight® per month (IU/kg BW/month) for prevention | Week 0- 104
Consumption of NovoEight® (IU/kg BW) from the day of surgery until the day of return to preventive regimen or on-demand treatment regimen | Week 0- 104

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry GCR, 1452, Study Director — Novo Nordisk A/S
Locations (2):
- Japan (2):
  - Novo Nordisk Investigational Site, Suginami-ku, Tokyo
  - Novo Nordisk Investigational Site, Tokyo

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com